CLINICAL TRIAL: NCT02265783
Title: Sensor Off Study Using a Nellcor USB Pulse Oximetry Monitor Interface Cable
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: COVMOPR0461
Record Dates: First submitted 2014-10-03; First posted 2014-10-16 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: Focus of Study: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nellcor USB Pulse Oximeter Monitor Interface Cable Sensor Test (Other)
  Interventions: Device: Nellcor USB Pulse Oximeter Monitor Interface Cable

INTERVENTIONS:
Device: Nellcor USB Pulse Oximeter Monitor Interface Cable — Volunteers are subjected to certain simulated, sensor removal conditions known to represent challenges to the sensor-off feature. Such conditions include exposing the sensor to an ambient light source, sensor slipping off the finger with the light emitter and detector facing each other or a sensor slipping off under a blanket.

SUMMARY:
The purpose of this study is to validate that the device posts a Sensor-Off message within the time frame stated in the proposed claims.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 or older (inclusive)
* Subject is able to participate for the duration of the study
* Subject is willing to sign an informed consent

Exclusion Criteria:

* Previous injury or trauma to fingers or hands that may change blood flow or vascular supply and affect our ability to test sensors
* Physiologic abnormalities that prevent proper application of pulse oximetry sensor
* Severe contact allergies that cause a reaction to standard adhesive materials such as those found in medical sensors and electrodes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Heyer, MD, Principal Investigator — Medtronic - MITG
Locations (1):
- Boulder Clinical Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The data will not be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- The Oxicable Pulse Oximetry Device: The subjects sit in a chair while a pulse oximetry sensor, hooked to the Oxicable pulse oximeter and a data collection system, is placed and removed in a certain sequence. This is done to demonstrate that the sensor-off feature displays per specifications when subjected to certain simulated, sensor removal conditions known to represent challenges to the sensor-off feature.
Period: Overall Study
Arm/Group | The Oxicable Pulse Oximetry Device
Started | 20
Completed | 20 (All subjects completed, one excluded from the analysis due to an issue with the data collection)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | The Oxicable Pulse Oximetry Device
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Report the Time Until the Device Posts "Sensor Off" After the Sensor is Removed
Description: A series of sensor-off events were collected from subjects in the study using marketed, off-the-shelf sensors. Each event was marked as pass if event duration (Timeend - Timestart) was less than or equal to 60 seconds; otherwise, the event was marked as greater than or equal to 60 seconds. The acceptance criteria is if 90% of the time the product posts Sensor Off, or any equal or higher priority alarm, within 60 seconds after sensor is removed.
Time Frame: 1 minute per event, multiple events per subject. Total duration up to 1 hour
Population: 20 subjects participated. There were errors with the data collection device for one subject and the data was unusable.
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | The Oxicable Pulse Oximetry Device
Number analyzed (Participants) | 19
Percent | 98.7 [96.2 to 100]

ADVERSE EVENTS:
Arm/Group | The Oxicable Pulse Oximetry Device
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No